CLINICAL TRIAL: NCT03601338
Title: Second Generation Low Molecular Weight Heparin (Bemiparin) as a Prophylactic for Management of Subsequent Pregnancy After an Unexplained Stillbirth: A Clinical Comparative Study
Brief Title: Low Molecular Weight Heparin in Pregnancies With Unexplained Stillbirths
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Shahla Alalaf, professor, Hawler Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HawlerMU2.7
Record Dates: First submitted 2018-07-18; First posted 2018-07-26 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Unexplained Stillbirth
Keywords: Unexplained stillbirth; Low molecular Weight Heparin; Umbilical artery; Doppler Ultrasound; Antenatal care
MeSH Terms: interventions — bemiparin; Geritol

STUDY DESIGN:
Intervention Model Description: pregnant women with history of unexplained fetal death
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bemiparin group (Active Comparator): Women with high resistant index of umbilical artery received the intervention Bemiparin Sodium 2,500 IU anti Xa/0.2 ml solution for injection in pre-filled syringe provided for each woman . The injections were received daily since 20 weeks gestation and up to 24 hours before delivery
  Other Name: Hibor; Laboratories Rovi pharmaceuticals
  Interventions: Drug: Bemiparin
- control group (Placebo Comparator): Normal umbilical arty resistant index group received only multivitamins and routine antenatal follow up
  Interventions: Other: multivitamins and routine antenatal follow up

INTERVENTIONS:
Drug: Bemiparin — second generation low molecular weight Heparin
  Other Names: Hibor
  Arms: Bemiparin group
Other: multivitamins and routine antenatal follow up — multivitamins and routine antenatal follow up
  Arms: control group

SUMMARY:
Bemiparin for pregnant women with abnormal umbilical artery Doppler ultrasound

DETAILED DESCRIPTION:
152 women with history of unexplained stillbirths were identified , umbilical arty Doppler ultrasound was conducted for them at 20-22 weeks gestation . they were divided into two group , group one are those with abnormal resistant index (= or more than 0.6) thy received Bemiparin 2500 IU subcutaneously daily up to 24 hours before delivery .

Group 2 with normal umbilical artery resistant index received no any interventions just routine antenatal follow up .

ELIGIBILITY:
Inclusion Criteria:

* Second pregnancy after previous unexplained fetal death
* Singleton pregnancy
* No any medical disorders during pregnancy like diabetes or Systemic Lupus Erythematosus
* Normally located placenta
* No congenital fetal anomalies
* Patient accept to participate

Exclusion Criteria:

* Confirmed thrombophilia
* Twin pregnancies
* Refused to participate

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-06 (Actual)

PRIMARY OUTCOMES:
Stillbirth | after 20 weeks gestation to the delivery of fetus
  Intrauterine fetal death
Early neonatal death | First week of life
  Death of newborn
Low birth weight | first hour of life
  New borne with birth weight less than 5th percentile in kilogram

SECONDARY OUTCOMES:
Preterm labor | 20-37 weeks
  delivery of the fetus before 37 weeks gestation
Pre-eclampsia | 20-41 week gestation
  High blood pressure with protein urea
major abruptio placenta | 20-41 week gestation
  Antepartum hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: shahla k. Alalaf, M.D, Principal Investigator — Hawler Medical University, college of Medicine, department of Obstetrics and Gynecology; Ariana K. Jawad, CABOG, Study Director — Kurdistan Board for Medical Specialist; Mahabad S. Ali, Diploma, Study Chair — Maternity Teaching Hospital
Locations (1):
- Hawler Medical University, Erbil, Kurdistan Region, Iraq